CLINICAL TRIAL: NCT03365167
Title: Clinical Evaluation of the Effect of LANAP (Laser Assisted New Attachment Procedure) as an Adjunct Treatment in Management of Patients With Chronic Periodontitis( Randomized Clinical Trial Study)
Brief Title: Clinical Evaluation of the Effect of LANAP as an Adjunct Treatment in Management of Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Neda Moslemi, Associate professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 96-02-97-36092
Record Dates: First submitted 2017-10-25; First posted 2017-12-07 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Periodontitis; Laser
Keywords: LANAP; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LANAP (Active Comparator): LANAP (Laser Assisted New Attachment Procedure)
  Interventions: Radiation: LANAP (Laser Assisted New Attachment Procedure)
- LANAP off (Placebo Comparator): laser therapy in off mode
  Interventions: Radiation: LANAP off

INTERVENTIONS:
Radiation: LANAP (Laser Assisted New Attachment Procedure) — radiation of Nd:YAG laser in periodontal pocket
  Arms: LANAP
Radiation: LANAP off — radiation of Nd:YAG laser in off mode in periodontal pocket
  Arms: LANAP off

SUMMARY:
this study evaluate the effect of LANAP (Laser Assisted New Attachment Procedure) as an Adjunct Treatment in Management of Patients With Chronic Periodontitis and assay the effect of LANAP on periodontal indexes like BOP, CAL, probing depth

DETAILED DESCRIPTION:
this study evaluate the effect of LANAP (Laser Assisted New Attachment Procedure) as an Adjunct Treatment in Management of Patients With Chronic Periodontitis and assay the effect of LANAP on periodontal indexes like BOP, CAL, probing depth in a split mouth design before treatment and after follow up sessions.

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of chronic periodontitis with at least two teeth with periodontal pocket depth more than 4 mm in each side

Exclusion Criteria:

* pregnant smoker systemic disease breast feeding

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
change of periodontal pocket depth | 0,1,2,3,4,5,6 months
  depth of periodontal pocket of each tooth

SECONDARY OUTCOMES:
change of Bleeding on Probing | 0,1,2,3,4,5,6 month
  sign of bleeding after 1 minutes post probing the tooth pocket
change of Full Mouth Bleeding Score | 0,1,2,3,4,5,6 month
  Bleeding Score of all teeth that is calculated by counting the Four dental levels that have sign of bleeding post probing (including , mesio-buccal,mid- buccal, disto-buccal and lingual) divided by the total number of total teeth in the mouth *4
change of Clinical attachment loss | 0,1,2,3,4,5,6 month
  distance from depth of tooth sulcus to cemento-enamel junction
change of Full Mouth Plaque Score | 0,1,2,3,4,5,6 month
  the number of 4 surfaces of each tooth(mesiobuccal, mid buccal, disto buccal and lingual surfaces) that have plaque that is disclosed by disclosing tables , then counting the number of the colored surface of all teeth divided by the total number of total teeth in the mouth*4

CONTACTS AND LOCATIONS:
Locations (1):
- Neda Moslemi, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dortaj D, Bassir SH, Hakimiha N, Hong H, Aslroosta H, Fekrazad R, Moslemi N. Efficacy of Nd:YAG laser-assisted periodontal therapy for the management of periodontitis: A double-blind split-mouth randomized controlled clinical trial. J Periodontol. 2022 May;93(5):662-672. doi: 10.1002/JPER.21-0242. Epub 2021 Sep 12. PMID 34411291